CLINICAL TRIAL: NCT03360630
Title: Autologous Dendritic Cell-cytokine Induced Killer Cell Immunotherapy Combined Anti-PD1 in Advanced NSCLC: A Randomized Controlled Trial
Brief Title: Anti-PD-1 Alone or Combined With Autologous Cell Therapy in Advanced NSCLC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: Duke University (Other); Geneplus-Beijing Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Jun Ren MD, PhD, Director, Comprehensive Cancer Center, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PD-1 plus DC-CIK for NSCLC
Record Dates: First submitted 2017-11-27; First posted 2017-12-04 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Lung Cancer; Neoplasms
MeSH Terms: conditions — Lung Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-PD-1 plus DC-CIK (Experimental)
  Interventions: Biological: Anti-PD-1 plus DC-CIK
- Anti-PD-1 alone (Active Comparator)
  Interventions: Biological: Anti-PD-1 alone

INTERVENTIONS:
Biological: Anti-PD-1 plus DC-CIK — Patients will receive pembrolizumab 100mg every three weeks until disease progression, unacceptable toxicity or patient refusal. DC-CIK Immunotherapy: Mononuclear cells were collected aseptically with blood cell separator composition apheresis, and cultured DC-CIK cells for 10-14 days. Cells were infused back to the patients in 3 times via intravenous infusion .Patients will received at least 2 cycles of DC-CIK Immunotherapy along with 4 dosage of anti-PD-1 antibody treatment. If the evaluation of the treatment is partial response or stable disease, additional cycles were eligible.
  Arms: Anti-PD-1 plus DC-CIK
Biological: Anti-PD-1 alone — Patients will receive pembrolizumab 100mg every three weeks until disease progression, unacceptable toxicity or patient refusal.
  Arms: Anti-PD-1 alone

SUMMARY:
A randomized controlled study to compared the clinical effects and safety of immunotherapy with dendritic cells and cytokine-induced killer cells administered with anti-PD-1 antibody in advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced or metastatic NSCLC.
* Patients must have received previously standard therapy for that malignancy or declined to chemotherapy/radiotherapy.
* Estimated life expectancy > 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0,1 or 2.
* Age 18 to 80.
* Adequate hematologic function, with WBC ≥ 3000/microliter, hemoglobin ≥ 9 g/dL (it is acceptable to have had prior transfusion), platelets ≥ 75,000/microliter; PT-INR <1.5 (unless patient is receiving warfarin in which case PT-INR must be <3), PTT <1.5X ULN
* Adequate renal and hepatic function, with serum creatinine < 1.5 mg/ dL, bilirubin < 1.5 mg/dL (except for Gilbert's syndrome which will allow bilirubin ≤ 2.0 mg/dL), ALT and AST ≤ 2.5 x upper limit of normal.

Exclusion Criteria:

* Patients with a history of autoimmune disease, such as but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis. Autoimmune related thyroid disease and vitiligo are permitted.
* Patients with serious intercurrent chronic or acute illness, such as cardiac disease (NYHA class III or IV), hepatic disease, or other illness considered by the Principal Investigator as unwarranted high risk for investigational drug treatment.
* Patients with a medical or psychological impediment to probable compliance with the protocol should be excluded.
* Concurrent (or within the last 5 years) second malignancy other than non melanoma skin cancer, cervical carcinoma in situ, controlled superficial bladder cancer, or other carcinoma in situ that has been treated.
* Presence of an active acute or chronic infection including: a urinary tract infection, HIV (as determined by ELISA and confirmed by Western Blot). Patients with HIV are excluded based on immuno-suppression, which may render them unable to respond to the vaccine; patients with chronic hepatitis are excluded because of concern that hepatitis could be exacerbated by the injections.
* Patients on chronic steroid therapy (or other immuno-suppressives, such as azathioprine or cyclosporin A) are excluded on the basis of potential immune suppression. Patients must have had 6 weeks of discontinuation of any steroid therapy (except that used as pre-medication for chemotherapy or contrast-enhanced studies or for acute treatment (<5 days) of intercurrent medical condition such as a gout flare) prior to enrollment.
* Pregnant and nursing women should be excluded from the protocol since this research may have unknown and harmful effects on an unborn child or on young children. If the patient is sexually active, the patient must agree to use a medically acceptable form of birth control while receiving treatment and for a period of 4 months following the last vaccination therapy. It is not known whether the treatment used in this study could affect the sperm and could potentially harm a child that may be fathered while on this study.
* Patients with acute or chronic skin disorders that will interfere with injection into the skin of the extremities or subsequent assessment of potential skin reactions will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival of the participants | 12 months
  From starting date of anti-PD-1 antibody treatment until date of until the date of first documented disease progression or date of death from any cause, whichever comes first.

SECONDARY OUTCOMES:
Overall survival of the participants(OS) | 24 months
  From starting date of anti-PD-1 antibody treatment until date of death from any cause
Assessment of Patient- Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PROCTCAE) | 24 months
  To assess and compare the PRO-CTCAE by patients receiving immunotherapy
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 24 months
Molecular Tumor Burden Index | 24 months
  Using mutation detection in ctDNA by liquid biopsy to assess tumor dynamics

OTHER OUTCOMES:
Cell-free tumor DNA | 24 months
  To investigate the relationship of ctDNA with clincial outcomes
Tumor related antigen peptides | 24 months
  To investigate the relationship of tumor related antigen peptides with clincial outcomes
T cell metaboic activity | 24 months
  To investigate the relationship of T cell metaboic activity with clincial outcomes
Microbial bacteria | 24 months
  To investigate the relationship of microbial bacteria with clincial outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Medical Unvierstiy Cancer Center/ Beijing Shijitan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No